CLINICAL TRIAL: NCT06963684
Title: Glaucoma Laser Assessment of Stability and Sustainability: Evaluating Long-Term Stability and Retreatment Efficacy of DSLT in Patients With Ocular Hypertension, Glaucoma Suspects, and Mild/Moderate POAG.
Brief Title: Glaucoma Laser Assessment of Stability and Sustainability
Acronym: GLASS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Twin Cities Eye Consultants (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCEC-003
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Glaucoma
Keywords: DSLT; glaucoma; IOP; intraocular pressure
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: All participants will receive DSLT treatment in both eyes at Baseline. 3-months later, one eye will be randomized to receive a second DSLT treatment. The primary endpoint is the difference in mean IOP between the dual-treatment and single-treatment eyes at 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental - Dual DSLT Treatment (Experimental): This study consists of a single arm using a paired-eye design. All participants will receive DSLT treatment in both eyes at Baseling. Then, one randomized eye receives a second DSLT treatment three months after the first.
  Interventions: Device: Dual-Treatment Direct Selective Laser Trabeculoplasty (DSLT)

INTERVENTIONS:
Device: Dual-Treatment Direct Selective Laser Trabeculoplasty (DSLT) — This is the first clinical study to evaluate repeat bilateral Direct Selective Laser Trabeculoplasty (DSLT) in treatment-naïve patients, using a paired-eye design. Unlike prior SLT studies, which focused on monocular treatment or repeat treatment following IOP rebound, this study randomizes one eye to receive a second DSLT treatment three months after the first, while the fellow eye receives only a single treatment. This allows for a direct intra-subject comparison of efficacy and durability. Existing studies, including GLAUrious and LiGHT, suggest the potential benefits of repeat laser, but no data currently exist for early, scheduled repeat treatment with DSLT. This trial uniquely investigates whether proactively repeating the procedure in a controlled eye extends IOP reduction and delays or reduces the need for topical medications.

SUMMARY:
The GLASS Study is designed to help researchers learn whether repeating a non-invasive laser treatment called DSLT (Direct Selective Laser Trabeculoplasty) can better control eye pressure in patients with early-stage glaucoma or ocular hypertension. All participants will receive the laser treatment in both eyes. After three months, one eye will be randomly selected to receive a second treatment, while the other eye will serve as a comparison. The goal is to see whether two treatments work better than one at keeping eye pressure low without using daily eye drops. This study will help doctors decide the best way to use this laser treatment to manage glaucoma and delay the need for medication. Participants will be followed for one year to monitor safety, eye pressure, and the need for any additional treatments.

DETAILED DESCRIPTION:
The GLASS Study (Glaucoma Laser Assessment of Sequential Sessions) is a prospective, interventional, paired-eye, single-site, investigator-initiated clinical trial designed to evaluate the safety and effectiveness of repeated applications of Direct Selective Laser Trabeculoplasty (DSLT) in treatment-naive patients with ocular hypertension (OHT), glaucoma suspect, or mild to moderate primary open-angle glaucoma (POAG).

DSLT is a non-contact, automated laser procedure that delivers 120 laser pulses evenly around the limbus to stimulate aqueous outflow by targeting the trabecular meshwork. The procedure is performed with the patient in an upright seated position using the Voyager DSLT device (Alcon). Unlike conventional SLT, this method does not require gonioscopy, coupling gel, or a contact lens.

All enrolled subjects must be treatment-naive, meaning they have not previously been on any ocular hypotensive medications. Eligible subjects will first complete a screening visit to verify inclusion and exclusion criteria. If criteria are met, they will be enrolled and proceed to the Baseline visit, where both eyes will undergo DSLT.

At the 3-month visit, one randomly selected eye (the "dual-treatment eye") will undergo a second DSLT session. The fellow eye (the "single-treatment eye") will receive no further laser treatment and serve as a control. Subjects will continue follow-up visits at 4 months (1 month after the second treatment), 6 months, 9 months, and 12 months from the baseline treatment.

Each study visit will include assessments such as best-corrected visual acuity (BCVA), intraocular pressure (IOP) via Goldmann applanation tonometry, slit-lamp examination, adverse event monitoring, ocular medication review (if applicable), and specular microscopy to assess corneal endothelial cell density. The primary endpoint is the difference in mean IOP between the dual-treatment and single-treatment eyes at 12 months.

Secondary endpoints include change in IOP from baseline at each follow-up timepoint, time to re-initiation of ocular hypotensive medications, and any difference in safety or complication rates between the two eyes.

The hypothesis is that a second treatment at the 3-month mark will provide enhanced and more durable IOP reduction, possibly reducing or delaying the need for medication. While DSLT has been studied previously in single-treatment applications, this is the first prospective trial evaluating repeat bilateral DSLT in a paired-eye design using one eye as its own internal control.

All procedures will be conducted at Twin Cities Eye Consultants in Minnesota. The study is sponsored and monitored internally by Twin Cities Eye Consultants' Research Committee, who will oversee compliance, data integrity, and protocol adherence.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 40 years or older
* A bilateral diagnosis of ocular hypertension, glaucoma suspect, or mild primary open angle glaucoma as defined by AAO PPP
* Treatment naïve with an unmedicated IOP between 21-35 mmHg, inclusive, and within +/- 3mmHg of each eye to be eligible
* BCVA of 20/50 or better
* The subject is able to read and understand the requirements of the study and provide written informed consent.
* The subject is willing to follow study instructions, agrees to comply with all study procedures and attend all scheduled follow-up exams for 12 months after the initial treatment.

Exclusion Criteria:

* Unable to view scleral spur inferiorly with gonioscopy.
* Congenital or developmental glaucoma, angle closure glaucoma, secondary glaucoma (e.g. exfoliative, pigmentary, etc.) pigmentary, neovascular glaucoma, closed angle glaucoma, or uveitic glaucoma.
* Use of oral or ocular hypotensive medication for glaucoma.
* Prior history of ocular surgery except for cataract surgery (must be ≥ 2 years prior)
* Clinically significant ocular pathology, other than cataract and glaucoma, including but not limited to neovascular age-related macular degeneration, advanced dry macular degeneration, and proliferative diabetic retinopathy, etc.
* Clinically significant ocular inflammation or infection within 6 months prior to screening.
* Previous corneal transplant or clinically significant corneal dystrophy, e.g., Fuch's dystrophy (≥12 confluent guttae)
* Unclear ocular media prevent visualization of the fundus or anterior chamber angle.
* Uncontrolled systemic disease that in the opinion of the Investigator would put the subject's health at risk and/or prevent the subject from completing all study visits.
* Current participation in another investigational drug or device clinical trial (which includes the fellow eye) within the past 30 calendar days.
* Pregnant or nursing women; or women of childbearing age not using medically acceptable contraceptives.

Accepted prior ocular procedures:

* Cataract surgery (if ≥ 2 years or screening)
* YAG capsulotomy (if ≥ 60 days of screening)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Mean Decrease in Intraocular Pressure (IOP) from Baseline | Baseline to Month 3
  Mean IOP reduction from untreated baseline (T0) to 3 months following bilateral DSLT, averaged between both eyes at the two timepoints.

SECONDARY OUTCOMES:
Mean IOP at 6 Months Post-DSLT Initiation | Month 6
  Comparison of mean IOP between the once-treated eye and the twice-treated eye at 6 months.
Proportion of Eyes Requiring No Additional Treatment | Month 6 and Month 12
  Proportion of eyes that remain drop-free and do not require additional glaucoma treatment at 6 and 12 months, comparing once- vs. twice-treated eyes.
Mean IOP at 12 Months Post-DSLT Initiation | Month 12
  Comparison of mean IOP between the once-treated eye and the twice-treated eye at 12 months.
Mean Percent Reduction in IOP from Baseline | Month 6 and Month 12
  Mean percentage reduction in IOP from baseline to 6 and 12 months, comparing once- vs. twice-treated eyes.

OTHER OUTCOMES:
Change in Conjunctival and Corneal Staining for Limbal Stem Cell Deficiency | Month 3 and Month 12
  Evaluation of conjunctival and corneal staining scores (0=no staining, 4=significant staining) to detect potential signs of limbal stem cell deficiency over the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: George R Wandling, MD, Principal Investigator — Twin Cities Eye Consultants - Partner
Locations (1):
- Twin Cities Eye Consultants, Coon Rapids, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo, Y., Ioannidou, A., & Jute, P. (2019). Selective laser trabeculoplasty: a review of repeatability. Annals Of Eye Science, 4(4), 20. doi:10.21037/aes.2019.05.01
- [Background] Polat J, Grantham L, Mitchell K, Realini T. Repeatability of selective laser trabeculoplasty. Br J Ophthalmol. 2016 Oct;100(10):1437-41. doi: 10.1136/bjophthalmol-2015-307486. Epub 2016 Feb 1. PMID 26834070
- [Background] Durr GM, Harasymowycz P. The effect of repeat 360-degree selective laser trabeculoplasty on intraocular pressure control in open-angle glaucoma. J Fr Ophtalmol. 2016 Mar;39(3):261-4. doi: 10.1016/j.jfo.2015.10.008. Epub 2016 Mar 16. PMID 26995075
- [Background] Jang HJ, Yu B, Hodge W, Malvankar-Mehta MS. Repeat Selective Laser Trabeculoplasty for Glaucoma Patients: A Systematic Review and Meta-analysis. J Curr Glaucoma Pract. 2021 Sep-Dec;15(3):117-124. doi: 10.5005/jp-journals-10078-1302. PMID 35173393